CLINICAL TRIAL: NCT01313312
Title: A Phase III, Multicentre, Prospective, Open Label Extension Study to Assess the Long Term Safety and Efficacy of Repeated Treatment of Dysport® Intramuscular Injections Used for the Treatment of Upper Limb Spasticity in Adult Subjects With Spastic Hemiparesis Due to Stroke or Traumatic Brain Injury
Brief Title: Dysport® Adult Upper Limb Spasticity Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y-52-52120-148; 2010-019162-83 (EudraCT Number)
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Nervous System Disorders
MeSH Terms: conditions — Nervous System Diseases | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Total Dysport® (Experimental): A total of 254 subjects in the open label study received between 1 and 5 intramuscular (i.m) injections of Dysport® according to their individual needs, for a period of up to 12 months. All subjects were administered an appropriate dosage of Dysport® (1000 Units [U] or 500 U) on Day 1 of treatment Cycle 1. At each study visit from Week 12 onwards, subjects were assessed to determine whether a subsequent treatment cycle was required and treatment cycles were administered at intervals of a minimum of 12 weeks apart depending on the subject's safety and efficacy response. From Cycle 2 onwards, a total dose of 1500 U could be administered in subjects requiring treatment with Dysport® in their shoulder and other upper limb muscles. Subjects who showed improvement in their upper limb during the first two treatment cycles were able to receive concomitant injections of Dysport® 500 U into at least one calf muscle, from Cycle 3 onwards as long as the total dose did not exceed 1500 U.
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A — Dysport® was supplied to the study centres in vials containing 500 U of botulinum toxin type A (BTX-A). Depending on the dose administered up to 3 vials were required for the injection.
  Each vial was reconstituted with sodium chloride for injection (0.9%). A total volume of 5.0 mL of the reconstituted product was injected for Dysport® 500 U and 1000 U, and 7.5 mL was injected for Dysport® 1500 U.
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The purpose of this research study is to assess the long term safety of Dysport® in hemiparetic subjects with upper limb spasticity due to stroke or traumatic brain injury over repeated treatment cycles.

DETAILED DESCRIPTION:
This was a phase III, multicentre, prospective, open label, repeat treatment cycles, extension to the double study Y-52-52120-145 (Study 145) . The study included both rollover subjects from Study 145 and de novo subjects. The primary study objective was to assess the long term safety of Dysport® in hemiparetic subjects with upper limb spasticity due to stroke or traumatic brain injury over repeated treatment cycles. The secondary study objective was to assess the long term efficacy of repeated treatment with Dysport®.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the double blind study, Y-52-52120-145

Exclusion Criteria:

* Major limitation in the passive range of motion in upper limb

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (34):
- United States (13):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - Associated Neurologist of Southern CT, PT, Fairfield, Connecticut
  - Parkinson's Disease & Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Design Neuroscience Miami, South Miami, Florida
  - The Rehabilitation Institute of Chicago, Chicago, Illinois
  - Mount Sinai School of Medicine, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Univ of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Medical Center, Winston-Salem, North Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Southwestern Medical Center at Dallas University of Texas, Dallas, Texas
  - University of North Texas HSC at Ben Hogan Center, Fort Worth, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah
- Belgium (2):
  - Université catholique de Louvain av Hippocrate 10, Brussels
  - Clinique Universitaire, Yvoir
- Charles University in Prague, Prague, Czechia
- France (7):
  - CHU Brest, Brest
  - Centre de Réadaptation de Coubert, Coubert
  - Centre Hospitalier Albert Chenevier-Hopital Henri Mondor, Créteil
  - Hopital Raymond Poincarré, Garches
  - Hôpital Sébastopol, Reims
  - CHU Strasbourg, Strasbourg
  - Hopital Rangueil, Toulouse
- Hungary (2):
  - Petz Aladar County Hospital, Gyor, Budapest
  - National Institute for Medical Rehabilitation, Budapest
- Italy (2):
  - Azienda Hospedaliero, Catania
  - Policlinico Universitario Agostino Gemelli, Roma
- Poland (3):
  - Malopolskie Centrum Medyczne, Krakow
  - Krakowska Akademia Neurologii, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
- Russia (3):
  - Medical Rehabilitation Center, Moscow
  - Scientific Center of Neurology of RAMS, Moscow
  - State University, Saint Petersburg
- Derer's Hospital, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Derived] Delafont B, Carroll K, Vilain C, Pham E. Investigation of mixed model repeated measures analyses and non-linear random coefficient models in the context of long-term efficacy data. Pharm Stat. 2018 Sep;17(5):515-526. doi: 10.1002/pst.1868. Epub 2018 May 20. PMID 29781237

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed as a multicentre study and included a total of 34 investigational sites in Belgium, the Czech Republic, France, Hungary, Italy, Poland, Russia, Slovakia and the United States of America (US) that included at least one subject. This study was an open label extension to the double blind Study 145 (Y-52-52120-145).
Pre-assignment Details: Of 227 subjects who completed Study 145, 4 subjects entered an observational phase and never received treatment with Dysport® in this open label extension study (Study 148). The remaining 223 subjects were eligible for retreatment and progressed to Study 148. In addition, 31 of the 34 de novo subjects screened were included in this study.
Groups:
- Total Dysport®: A total of 254 subjects in the open label study received between 1 and 5 intramuscular (i.m.) injections of Dysport® according to their individual needs, for a period of up to 12 months.
  All subjects were administered an appropriate dosage of Dysport® (1000 U or 500 U) on Day 1 of treatment Cycle 1. At each study visit from Week 12 onwards, subjects were assessed to determine whether a subsequent treatment cycle was required and treatment cycles were administered at intervals of a minimum of 12 weeks apart depending on the subject's safety and efficacy response.
  From Cycle 2 onwards, a total dose of 1500 U could be administered in subjects requiring treatment with Dysport® in their shoulder and other upper limb muscles. Subjects who showed improvement in their upper limb during the first two treatment cycles were able to receive concomitant injections of Dysport® 500 U into at least one calf muscle, from Cycle 3 onwards as long as the total dose did not exceed 1500 U.
Period: Overall Study
Arm/Group | Total Dysport®
Started | 258
Cycle 1 | 254
Cycle 2 | 229
Cycle 3 | 175
Cycle 4 | 81
Cycle 5 | 11
Completed | 222
Not Completed | 36
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 18
Not completed — Lack of Efficacy | 3
Not completed — Investigator Decision | 1
Not completed — Observational Phase | 1
Not completed — Subject Withdrawn Early in Error | 4
Not completed — Did Not Receive Treatment with Dysport® | 4

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the 254 Subjects who entered this open label study (223 from Study 145 and 31 de novo subjects) and received at least one open label injection of Dysport®.
Groups:
- Total Dysport®: A total of 254 subjects in the open label study received between 1 and 5 i.m. injections of Dysport® according to their individual needs, for a period of up to 12 months.
  All subjects were administered an appropriate dosage of Dysport® (1000 U or 500 U) on Day 1 of treatment Cycle 1. At each study visit from Week 12 onwards, subjects were assessed to determine whether a subsequent treatment cycle was required and treatment cycles were administered at intervals of a minimum of 12 weeks apart depending on the subject's safety and efficacy response.
  From Cycle 2 onwards, a total dose of 1500 U could be administered in subjects requiring treatment with Dysport® in their shoulder and other upper limb muscles. Subjects who showed improvement in their upper limb during the first two treatment cycles were able to receive concomitant injections of Dysport® 500 U into at least one calf muscle, from Cycle 3 onwards as long as the total dose did not exceed 1500 U.
Arm/Group | Total Dysport®
Number analyzed (Participants) | 254
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 201
  >=65 years | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 238
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 27
  White | 218
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Long-term Safety of Dysport® Through the Collection of Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE was reported as emergent if it arose (i.e. started or worsened in severity) in the treatment phase after the subject received study medication. Adverse events of special interest (AESIs) were identified as those assessed as being due to remote spread of effect of Dysport®, or any adverse event (AE) that was assessed as a hypersensitivity reaction. TEAEs, AESIs, severe TEAEs, serious adverse events (SAEs), treatment related TEAEs, TEAEs leading to withdrawal and fatal SAEs are summarised by treatment cycle.
Time Frame: Up to Week 52
Population: Subjects who entered the study and received at least one open label injection of Dysport® were evaluated for safety analysis. Only subjects with data available for analysis at the point of testing are reported.
Measure: Number; unit: Participants
Arm/Group | Total Dysport®
Number analyzed (Participants) | 254
Participants
  TEAEs: Cycle 1 | 102
  TEAEs: Cycle 2: number analyzed (Participants) | 229
  TEAEs: Cycle 2 | 62
  TEAEs: Cycle 3: number analyzed (Participants) | 175
  TEAEs: Cycle 3 | 47
  TEAEs: Cycle 4: number analyzed (Participants) | 81
  TEAEs: Cycle 4 | 11
  TEAEs: Cycle 5: number analyzed (Participants) | 11
  TEAEs: Cycle 5 | 2
  Treatment related TEAE: Cycle 1 | 18
  Treatment related TEAE: Cycle 2: number analyzed (Participants) | 229
  Treatment related TEAE: Cycle 2 | 8
  Treatment related TEAE: Cycle 3: number analyzed (Participants) | 175
  Treatment related TEAE: Cycle 3 | 5
  Treatment related TEAE: Cycle 4: number analyzed (Participants) | 81
  Treatment related TEAE: Cycle 4 | 2
  Treatment related TEAE: Cycle 5: number analyzed (Participants) | 11
  Treatment related TEAE: Cycle 5 | 0
  Severe TEAEs: Cycle 1 | 14
  Severe TEAEs: Cycle 2: number analyzed (Participants) | 229
  Severe TEAEs: Cycle 2 | 8
  Severe TEAEs: Cycle 3: number analyzed (Participants) | 175
  Severe TEAEs: Cycle 3 | 4
  Severe TEAEs: Cycle 4: number analyzed (Participants) | 81
  Severe TEAEs: Cycle 4 | 1
  Severe TEAEs: Cycle 5: number analyzed (Participants) | 11
  Severe TEAEs: Cycle 5 | 0
  TEAEs Leading to Withdrawal: Cycle 1 | 2
  TEAEs Leading to Withdrawal: Cycle 2: number analyzed (Participants) | 229
  TEAEs Leading to Withdrawal: Cycle 2 | 1
  TEAEs Leading to Withdrawal: Cycle 3: number analyzed (Participants) | 175
  TEAEs Leading to Withdrawal: Cycle 3 | 2
  TEAEs Leading to Withdrawal: Cycle 4: number analyzed (Participants) | 81
  TEAEs Leading to Withdrawal: Cycle 4 | 0
  TEAEs Leading to Withdrawal: Cycle 5: number analyzed (Participants) | 11
  TEAEs Leading to Withdrawal: Cycle 5 | 0
  AESIs: Cycle 1 | 2
  AESIs: Cycle 2: number analyzed (Participants) | 229
  AESIs: Cycle 2 | 0
  AESIs: Cycle 3: number analyzed (Participants) | 175
  AESIs: Cycle 3 | 0
  AESIs: Cycle 4: number analyzed (Participants) | 81
  AESIs: Cycle 4 | 0
  AESIs: Cycle 5: number analyzed (Participants) | 11
  AESIs: Cycle 5 | 0
  SAEs: Cycle 1 | 10
  SAEs: Cycle 2: number analyzed (Participants) | 229
  SAEs: Cycle 2 | 6
  SAEs: Cycle 3: number analyzed (Participants) | 175
  SAEs: Cycle 3 | 6
  SAEs: Cycle 4: number analyzed (Participants) | 81
  SAEs: Cycle 4 | 1
  SAEs: Cycle 5: number analyzed (Participants) | 11
  SAEs: Cycle 5 | 0
  Fatal SAEs: Cycle 1 | 1
  Fatal SAEs: Cycle 2: number analyzed (Participants) | 229
  Fatal SAEs: Cycle 2 | 1
  Fatal SAEs: Cycle 3: number analyzed (Participants) | 175
  Fatal SAEs: Cycle 3 | 1
  Fatal SAEs: Cycle 4: number analyzed (Participants) | 81
  Fatal SAEs: Cycle 4 | 0
  Fatal SAEs: Cycle 5: number analyzed (Participants) | 11
  Fatal SAEs: Cycle 5 | 0

2. Primary Outcome: Mean Change From Baseline to End of Study/Early Withdrawal in Diastolic and Systolic Blood Pressure (BP)
Description: Systolic and diastolic BP were recorded at screening, baseline and at each post baseline visit. Vital signs were measured with the subject in a sitting position after resting for 3 minutes. Outcome measure is reported for number of subjects with data available for analysis.
Time Frame: Up to Week 52
Population: as for outcome 1
Measure: Mean (Full Range); unit: Millimeters of Mercury (mm Hg)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 238
Millimeters of Mercury (mm Hg)
  Diastolic BP | 0 [-29 to 34]
  Systolic BP | -2.8 [-63 to 41]

3. Primary Outcome: Mean Change From Baseline to End of Study/Early Withdrawal in Heart Rate (HR)
Description: HR was recorded at screening, baseline and at each post baseline visit. Vital signs were measured with the subject in a sitting position after resting for 3 minutes. Outcome measure is reported for number of subjects with data available for analysis.
Time Frame: Up to Week 52
Population: as for outcome 1
Measure: Mean (Full Range); unit: Beats per minute (bpm)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 239
Beats per minute (bpm) | 2.5 [-28 to 30]

4. Primary Outcome: Mean Change From Baseline to End of Study/Early Withdrawal in Red Blood Cell (RBC) Count
Description: Blood samples for RBC count were taken at baseline, at post treatment follow up visit Week 4, and at end of study/early withdrawal. Outcome measure is reported for number of subjects with data available for analysis.
Time Frame: Up to Week 52
Population: as for outcome 1
Measure: Mean (Full Range); unit: Tera cells/Litre (L)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 219
Tera cells/Litre (L) | 0.03 [-1.15 to 1.06]

5. Primary Outcome: Mean Change From Baseline to End of Study/Early Withdrawal in Haemoglobin and Mean Corpuscular Haemoglobin Concentration (MCHC)
Description: Blood samples for haemoglobin and MCHC were taken at baseline, at post treatment follow up visit Week 4, and at the end of study/early withdrawal. Outcome measure is reported for number of subjects with data available for analysis.
Time Frame: Up to Week 52
Population: as for outcome 1
Measure: Mean (Full Range); unit: grams(g)/L
Arm/Group | Total Dysport®
Number analyzed (Participants) | 219
grams(g)/L
  Haemoglobin | -0.7 [-33 to 37]
  MCHC | -0.8 [-26 to 34]

6. Primary Outcome: Mean Change From Baseline to End of Study/Early Withdrawal in Haematocrit
Description: Blood samples for haematocrit were taken at baseline, at post treatment follow up visit Week 4, and at end of study/early withdrawal. Outcome measure is reported for number of subjects with data available for analysis.
Time Frame: Up to Week 52
Population: as for outcome 1
Measure: Mean (Full Range); unit: percentage of RBC in blood
Arm/Group | Total Dysport®
Number analyzed (Participants) | 219
percentage of RBC in blood | -0.0011 [-0.104 to 0.087]

7. Primary Outcome: Mean Change From Baseline to End of Study/Early Withdrawal in Mean Corpuscular Haemoglobin (MCH)
Description: Blood samples for MCH were taken at baseline, at post treatment follow up visit Week 4, and at end of study/early withdrawal. Outcome measure is reported for number of subjects with data available for analysis.
Time Frame: Up to Week 52
Population: as for outcome 1
Measure: Mean (Full Range); unit: picograms (pg)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 219
picograms (pg) | -0.33 [-5 to 4.9]

8. Primary Outcome: Mean Change From Baseline to End of Study/Early Withdrawal in Mean Corpuscular Volume (MCV)
Description: Blood samples for MCV were taken at baseline, at post treatment follow up visit Week 4, and at end of study/early withdrawal. Outcome measure is reported for number of subjects with data available for analysis.
Time Frame: Up to Week 52
Population: as for outcome 1
Measure: Mean (Full Range); unit: femtoliters (fL)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 219
femtoliters (fL) | -0.77 [-9.9 to 8.2]

9. Primary Outcome: Mean Change From Baseline to End of Study/Early Withdrawal in White Blood Cell (WBC) Count, Neutrophils, Lymphocytes and Platelets
Description: Blood samples for WBC count with differentials (neutrophils, lymphocytes) and platelet count were taken at baseline, at post treatment follow up visit Week 4, and at end of study or early withdrawal.
Time Frame: Up to Week 52
Population: as for outcome 1
Measure: Mean (Full Range); unit: Giga cells/L
Arm/Group | Total Dysport®
Number analyzed (Participants) | 219
Giga cells/L
  WBC count | 0.04 [-6.5 to 5.2]
  Neutrophils | 0 [-6.8 to 5.6]
  Lymphocytes | 0.01 [-1.9 to 1.2]
  Platelets: number analyzed (Participants) | 214
  Platelets | 3.2 [-142 to 249]

10. Primary Outcome: Mean Change From Baseline to End of Study/Early Withdrawal in 12-Lead Electrocardiogram (ECG)
Description: 12-lead ECG tracing was performed at baseline, post treatment at Week 4 and at the end of study/early withdrawal visit. The 12-lead ECG recordings were performed at a paper speed of 25 mm/s, recorded with the subject in a supine position after 5 minutes rest. The ECG parameters reported were QRS duration, PR duration, QT duration, QTcB (QT interval corrected for HR according to Bazett), and QTcF (QT interval corrected for HR according to Fridericia) at baseline and the change to end of study/early withdrawal visit (EOS).
Time Frame: Up to Week 52
Population: The ECG analysis was performed in the safety population among subjects who had at least one ECG measurement before injection and at least one ECG after injection. Only subjects with data available for analysis at the point of testing are reported.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 235
milliseconds (ms)
  QT Duration - Baseline: number analyzed (Participants) | 233
  QT Duration - Baseline | 403.6 (31.9)
  QT Duration - Change from Baseline to EOS: number analyzed (Participants) | 210
  QT Duration - Change from Baseline to EOS | -6.3 (22.1)
  QTcF - Baseline: number analyzed (Participants) | 233
  QTcF - Baseline | 417.8 (22.9)
  QTcF - Change from Baseline to EOS: number analyzed (Participants) | 210
  QTcF - Change from Baseline to EOS | -1 (15.5)
  QTcB - Baseline: number analyzed (Participants) | 233
  QTcB - Baseline | 425.6 (25.5)
  QTcB - Change from Baseline to EOS: number analyzed (Participants) | 210
  QTcB - Change from Baseline to EOS | 1.9 (20.2)
  QRS Duration - Baseline | 94.9 (15.3)
  QRS Duration - Change from Baseline to EOS: number analyzed (Participants) | 210
  QRS Duration - Change from Baseline to EOS | -0.4 (6.4)
  PR Duration - Baseline: number analyzed (Participants) | 233
  PR Duration - Baseline | 165.6 (25.4)
  PR Duration - Change from Baseline to EOS: number analyzed (Participants) | 210
  PR Duration - Change from Baseline to EOS | -0.3 (13.2)

11. Primary Outcome: Mean Change From Baseline to End of Study/Early Withdrawal in Alkaline Phosphatase (ALP), Gamma Glutamyl Transferase (GGT), Serum Glutamic Oxaloacetic Transaminase (SGOT) and Serum Glutamic Pyruvic Transaminase (SGPT)
Description: Blood samples for analysis of the following clinical chemistry parameters: ALP, GGT, SGOT and SGPT were taken at baseline, at post treatment follow up visit Week 4, and at end of study/early withdrawal. Outcome measure is reported for number of subjects with data available for analysis.
Time Frame: Up to Week 52
Population: as for outcome 1
Measure: Mean (Full Range); unit: International Unit/L (IU/L)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 226
International Unit/L (IU/L)
  ALP | -0.6 [-39 to 83]
  SGOT | 1.4 [-32 to 45]
  SGPT | 1.2 [-81 to 57]
  GGT | 1.5 [-105 to 195]

12. Primary Outcome: Mean Change From Baseline to End of Study/Early Withdrawal in Total Bilirubin and Creatinine
Description: Blood samples for clinical chemistry analysis of total bilirubin and creatinine were taken at baseline, at post treatment follow up visit Week 4, and at end of study/early withdrawal. Outcome measure is reported for number of subjects with data available for analysis.
Time Frame: Up to Week 52
Population: as for outcome 1
Measure: Mean (Full Range); unit: Micromole/L (μmol/L)
Arm/Group | Total Dysport®
Number analyzed (Participants) | 226
Micromole/L (μmol/L)
  Total Bilirubin | -0.27 [-18.7 to 12.2]
  Creatinine | -3.7 [-115 to 35]

13. Primary Outcome: Mean Change From Baseline to End of Study/Early Withdrawal in Blood Urea Nitrogen (BUN) and Fasting Blood Glucose
Description: Blood samples for analysis of BUN and fasting blood glucose levels were taken at baseline, at post treatment follow up visit Week 4, and at end of study/early withdrawal.
Time Frame: Up to Week 52
Population: as for outcome 1
Measure: Mean (Full Range); unit: millimoles(mmol)/L
Arm/Group | Total Dysport®
Number analyzed (Participants) | 226
millimoles(mmol)/L
  BUN | -0.033 [-12.85 to 8.93]
  Fasting Blood Glucose: number analyzed (Participants) | 101
  Fasting Blood Glucose | 0.132 [-3.66 to 7.94]

14. Primary Outcome: Mean Change From Baseline to End of Study/Early Withdrawal in 12 Lead ECG - HR
Description: HR was measured by 12-lead ECG tracing, performed at baseline, at post treatment follow up visit Week 4, and at the end of study or early withdrawal visit. The 12-lead ECG recordings were performed at a paper speed of 25 mm/s, recorded with the subject in a supine position after 5 minutes rest.
Time Frame: Up to Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Total Dysport®
Number analyzed (Participants) | 243
bpm
  Baseline | 68.2 (11.3)
  Change from Baseline to EOS: number analyzed (Participants) | 226
  Change from Baseline to EOS | 2.7 (10.5)

15. Primary Outcome: Number of Subjects With Botulinum Toxin A Binding and Neutralising Putative Antibodies
Description: Blood samples were collected at baseline, Week 4 of each cycle, and at the end of study/early withdrawal to test for the presence of Botulinum Toxin A Binding antibodies. Samples positive for the presence of binding antibodies were then analysed for the presence of neutralising putative antibodies. The number of subjects who were either positive (+ve) or negative (-ve) at baseline and then positive post baseline for binding or neutralising antibodies were reported.
Time Frame: Up to Week 52
Population: Binding and neutralising antibodies were evaluated at baseline for all 258 subjects (rollover and de novo) enrolled in Study 148. Only subjects with data available for analysis at the point of testing are reported.
Measure: Number; unit: Participants
Arm/Group | Total Dysport®
Number analyzed (Participants) | 258
Participants
  Binding +ve at baseline | 5
  Binding -ve at baseline & +ve post baseline: number analyzed (Participants) | 251
  Binding -ve at baseline & +ve post baseline | 20
  Neutralising +ve at baseline | 4
  Neutralising -ve at baseline & +ve post baseline: number analyzed (Participants) | 252
  Neutralising -ve at baseline & +ve post baseline | 11

16. Secondary Outcome: Mean Change From Baseline Modified Ashworth Scale (MAS) in the Overall Primary Targeted Muscle Group (PTMG) for Upper Limb at Week 4
Description: The clinical assessment of muscle tone was performed using the MAS. The MAS consists of 6 grades: 0, 1, 1+, 2, 3, or 4 that can be applied to muscles of both the upper and lower limbs. The MAS was applied by the rater by stretching the joint through its full available range over 1 second. The mean changes from baseline to Week 4 in MAS in the overall PTMG (finger, wrist or elbow flexors) are reported.
Time Frame: At Week 4
Population: The Intent-to-Treat (ITT) population was all enrolled subjects who received at least one injection of study medication in this open label extension study. Too few subjects were treated in Cycle 5 to allow direct comparisons with other cycles and are not reported. Only subjects with data available for analysis at the point of testing are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 252
units on a scale
  Cycle 1 | -1.4 (1.1)
  Cycle 2: number analyzed (Participants) | 226
  Cycle 2 | -1.6 (1.2)
  Cycle 3: number analyzed (Participants) | 163
  Cycle 3 | -1.5 (1.1)
  Cycle 4: number analyzed (Participants) | 80
  Cycle 4 | -1.4 (1.1)

17. Secondary Outcome: Percentage of Subjects With at Least 1 or 2 Grade Reduction in MAS for Overall PTMG
Description: The MAS consists of 6 grades: 0, 1, 1+, 2, 3, or 4 that can be applied to muscles of both the upper and lower limbs. The MAS was applied by the rater by stretching the joint through its full available range over 1 second. The percentage of subjects with at least a 1 grade reduction and at least a 2 grades reduction from baseline in mean MAS in the overall PTMG at Week 4 are reported.
Time Frame: At Week 4
Population: The ITT population was defined as all enrolled subjects who received at least one injection of study medication in this open label extension study. Too few subjects were treated in Cycle 5 to allow direct comparisons with other cycles and are not reported. Only subjects with data available for analysis at the point of testing are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Total Dysport®
Number analyzed (Participants) | 254
percentage of participants
  At least 1 grade reduction - Cycle 1 | 77.6
  At least 1 grade reduction - Cycle 2: number analyzed (Participants) | 229
  At least 1 grade reduction - Cycle 2 | 79.5
  At least 1 grade reduction - Cycle 3: number analyzed (Participants) | 175
  At least 1 grade reduction - Cycle 3 | 77.1
  At least 1 grade reduction - Cycle 4: number analyzed (Participants) | 81
  At least 1 grade reduction - Cycle 4 | 75.3
  At least 2 grades reduction - Cycle 1 | 42.1
  At least 2 grades reduction - Cycle 2: number analyzed (Participants) | 229
  At least 2 grades reduction - Cycle 2 | 48.0
  At least 2 grades reduction - Cycle 3: number analyzed (Participants) | 175
  At least 2 grades reduction - Cycle 3 | 44.6
  At least 2 grades reduction - Cycle 4: number analyzed (Participants) | 81
  At least 2 grades reduction - Cycle 4 | 37.0

18. Secondary Outcome: Mean Change From Baseline MAS in the Extrinsic Finger Flexors at Week 4
Description: The clinical assessment of muscle tone was performed using the MAS. The MAS consists of 6 grades: 0, 1, 1+, 2, 3, or 4 that can be applied to muscles of both the upper and lower limbs. The MAS was applied by the rater by stretching the joint through its full available range over 1 second. The mean changes from baseline to Week 4 in MAS in the extrinsic finger flexors are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 220
units on a scale
  Cycle 1 | -1.3 (1.1)
  Cycle 2: number analyzed (Participants) | 191
  Cycle 2 | -1.5 (1.2)
  Cycle 3: number analyzed (Participants) | 141
  Cycle 3 | -1.5 (1.3)
  Cycle 4: number analyzed (Participants) | 69
  Cycle 4 | -1.3 (1.2)

19. Secondary Outcome: Percentage of Subjects With at Least 1 or 2 Grade Reduction in MAS for Extrinsic Finger Flexors at Week 4
Description: The MAS consists of 6 grades: 0, 1, 1+, 2, 3, or 4 that can be applied to muscles of both the upper and lower limbs. The MAS was applied by the rater by stretching the joint through its full available range over 1 second. The percentage of subjects with at least a 1 grade reduction and at least a 2 grades reduction from baseline in mean MAS in the extrinsic finger flexors at Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Number; unit: percentage of subjects
Arm/Group | Total Dysport®
Number analyzed (Participants) | 145
percentage of subjects
  At least 1 Grade Reduction -Cycle 1 | 78.6
  At least 1 Grade Reduction -Cycle 2: number analyzed (Participants) | 134
  At least 1 Grade Reduction -Cycle 2 | 81.3
  At least 1 Grade Reduction -Cycle 3: number analyzed (Participants) | 105
  At least 1 Grade Reduction -Cycle 3 | 80
  At least 1 Grade Reduction -Cycle 4: number analyzed (Participants) | 56
  At least 1 Grade Reduction -Cycle 4 | 80.4
  At least 2 Grades Reduction -Cycle 1 | 44.1
  At least 2 Grades Reduction -Cycle 2: number analyzed (Participants) | 134
  At least 2 Grades Reduction -Cycle 2 | 49.3
  At least 2 Grades Reduction -Cycle 3: number analyzed (Participants) | 105
  At least 2 Grades Reduction -Cycle 3 | 49.5
  At least 2 Grades Reduction -Cycle 4: number analyzed (Participants) | 56
  At least 2 Grades Reduction -Cycle 4 | 37.5

20. Secondary Outcome: Mean Change From Baseline MAS in the Wrist Flexors at Week 4
Description: The clinical assessment of muscle tone was performed using the MAS. The MAS consists of 6 grades: 0, 1, 1+, 2, 3, or 4 that can be applied to muscles of both the upper and lower limbs. The MAS was applied by the rater by stretching the joint through its full available range over 1 second. The mean changes from baseline to Week 4 in MAS in the wrist flexors are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 169
units on a scale
  Cycle 1 | -1.5 (1.2)
  Cycle 2: number analyzed (Participants) | 159
  Cycle 2 | -1.6 (1.3)
  Cycle 3: number analyzed (Participants) | 104
  Cycle 3 | -1.6 (1.3)
  Cycle 4: number analyzed (Participants) | 51
  Cycle 4 | -1.5 (1.2)

21. Secondary Outcome: Percentage of Subjects With at Least 1 or 2 Grade Reduction in MAS for Wrist Flexors at Week 4
Description: The MAS consists of 6 grades: 0, 1, 1+, 2, 3, or 4 that can be applied to muscles of both the upper and lower limbs. The MAS was applied by the rater by stretching the joint through its full available range over 1 second. The percentage of subjects with at least a 1 grade reduction and at least a 2 grades reduction in mean MAS in the wrist flexors at Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Number; unit: percentage of subjects
Arm/Group | Total Dysport®
Number analyzed (Participants) | 40
percentage of subjects
  At least 1 Grade Reduction -Cycle 1 | 62.5
  At least 1 Grade Reduction -Cycle 2: number analyzed (Participants) | 35
  At least 1 Grade Reduction -Cycle 2 | 74.3
  At least 1 Grade Reduction -Cycle 3: number analyzed (Participants) | 23
  At least 1 Grade Reduction -Cycle 3 | 73.9
  At least 1 Grade Reduction -Cycle 4: number analyzed (Participants) | 10
  At least 1 Grade Reduction -Cycle 4 | 50
  At least 2 Grades Reduction -Cycle 1 | 47.5
  At least 2 Grades Reduction -Cycle 2: number analyzed (Participants) | 35
  At least 2 Grades Reduction -Cycle 2 | 54.3
  At least 2 Grades Reduction -Cycle 3: number analyzed (Participants) | 23
  At least 2 Grades Reduction -Cycle 3 | 47.8
  At least 2 Grades Reduction -Cycle 4: number analyzed (Participants) | 10
  At least 2 Grades Reduction -Cycle 4 | 30.0

22. Secondary Outcome: Mean Change From Baseline MAS in the Elbow Flexors at Week 4
Description: The clinical assessment of muscle tone was performed using the MAS. The MAS consists of 6 grades: 0, 1, 1+, 2, 3, or 4 that can be applied to muscles of both the upper and lower limbs. The MAS was applied by the rater by stretching the joint through its full available range over 1 second. The mean changes from baseline to Week 4 in MAS in the elbow flexors are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 179
units on a scale
  Cycle 1 | -1.0 (1.0)
  Cycle 2: number analyzed (Participants) | 163
  Cycle 2 | -1.1 (1.1)
  Cycle 3: number analyzed (Participants) | 119
  Cycle 3 | -1.1 (1.1)
  Cycle 4: number analyzed (Participants) | 48
  Cycle 4 | -0.8 (1.0)

23. Secondary Outcome: Percentage of Subjects With at Least 1 or 2 Grade Reduction in MAS for Elbow Flexors at Week 4
Description: The MAS consists of 6 grades: 0, 1, 1+, 2, 3, or 4 that can be applied to muscles of both the upper and lower limbs. The MAS was applied by the rater by stretching the joint through its full available range over 1 second. The percentage of subjects at least a 1 grade reduction and at least a 2 grades reduction from baseline in mean MAS in the elbow flexors at Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Number; unit: percentage of subjects
Arm/Group | Total Dysport®
Number analyzed (Participants) | 69
percentage of subjects
  At least 1 Grade Reduction -Cycle 1 | 84.1
  At least 1 Grade Reduction -Cycle 2: number analyzed (Participants) | 60
  At least 1 Grade Reduction -Cycle 2 | 78.3
  At least 1 Grade Reduction -Cycle 3: number analyzed (Participants) | 45
  At least 1 Grade Reduction -Cycle 3 | 75.6
  At least 1 Grade Reduction -Cycle 4: number analyzed (Participants) | 15
  At least 1 Grade Reduction -Cycle 4 | 73.3
  At least 2 Grades Reduction -Cycle 1 | 34.8
  At least 2 Grades Reduction -Cycle 2: number analyzed (Participants) | 60
  At least 2 Grades Reduction -Cycle 2 | 41.7
  At least 2 Grades Reduction -Cycle 3: number analyzed (Participants) | 45
  At least 2 Grades Reduction -Cycle 3 | 33.3
  At least 2 Grades Reduction -Cycle 4: number analyzed (Participants) | 15
  At least 2 Grades Reduction -Cycle 4 | 40.0

24. Secondary Outcome: Mean Change From Baseline MAS in the Shoulder Extensors at Week 4
Description: The clinical assessment of muscle tone was performed using the MAS. The MAS consists of 6 grades: 0, 1, 1+, 2, 3, or 4 that can be applied to muscles of both the upper and lower limbs. The MAS was applied by the rater by stretching the joint through its full available range over 1 second. The mean changes from baseline to Week 4 in MAS in the shoulder extensors are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 81
units on a scale
  Cycle 1: number analyzed (Participants) | 31
  Cycle 1 | -0.9 (1.1)
  Cycle 2: number analyzed (Participants) | 64
  Cycle 2 | -0.7 (0.9)
  Cycle 3: number analyzed (Participants) | 54
  Cycle 3 | -0.6 (1.0)
  Cycle 4 | -0.6 (0.8)

25. Secondary Outcome: Physician's Global Assessment (PGA) of Treatment Response at Week 4
Description: The PGA is a 9-point rating scale: -4=markedly worse, -3=much worse, -2=worse, -1=slightly worse, 0=no change, +1=slightly improved, +2=improved, +3=much improved, +4=markedly improved. An assessment of overall treatment response was conducted by the investigator and the mean PGA scores during long-term open label treatment with Dysport were reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 253
units on a scale
  Cycle 1 | 1.7 (1)
  Cycle 2: number analyzed (Participants) | 227
  Cycle 2 | 1.9 (1)
  Cycle 3: number analyzed (Participants) | 167
  Cycle 3 | 1.9 (1)
  Cycle 4: number analyzed (Participants) | 80
  Cycle 4 | 2 (0.9)

26. Secondary Outcome: Mean Change From Baseline in Disability Assessment Scale (DAS) Score for the Principal Target of Treatment (PTT) at Week 4
Description: At baseline the subject and investigator together selected one of the four DAS domains as the PTT. The selected domain was required to have a rating of moderate or severe (≥2) at baseline. The DAS is a 4-point scale, the extent of functional impairment in 4 functional domains (dressing, hygiene, limb position and pain) was rated as follows: 0=no disability, 1=mild disability (noticeable but does not interfere significantly with normal activities), 2=moderate disability (normal activities require increased effort and/or assistance) and 3=severe disability (normal activities limited). The mean changes in DAS at Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 252
units on a scale
  Cycle 1 | -0.9 (0.8)
  Cycle 2: number analyzed (Participants) | 226
  Cycle 2 | -1.1 (0.8)
  Cycle 3: number analyzed (Participants) | 166
  Cycle 3 | -1.1 (0.8)
  Cycle 4: number analyzed (Participants) | 80
  Cycle 4 | -1.1 (0.8)

27. Secondary Outcome: Percentage of Subjects With at Least 1 Grade Reduction in DAS for PTT at Week 4
Description: At baseline the subject and investigator together selected one of the four DAS domains as the PTT. The selected domain was required to have a rating of moderate or severe (≥2) at baseline. The DAS is a 4-point scale, the extent of functional impairment in 4 functional domains (dressing, hygiene, limb position and pain) was rated as follows: 0=no disability, 1=mild disability (noticeable but does not interfere significantly with normal activities), 2=moderate disability (normal activities require increased effort and/or assistance) and 3=severe disability (normal activities limited). The percentage of subjects with at least 1 grade reduction from baseline in DAS for PTT at Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Number; unit: Percentage of Subjects
Arm/Group | Total Dysport®
Number analyzed (Participants) | 254
Percentage of Subjects
  Cycle 1 | 68.5
  Cycle 2: number analyzed (Participants) | 229
  Cycle 2 | 75.1
  Cycle 3: number analyzed (Participants) | 175
  Cycle 3 | 73.7
  Cycle 4: number analyzed (Participants) | 81
  Cycle 4 | 74.1

28. Secondary Outcome: Percentage of Subjects With at Least One Grade Reduction in DAS for Individual Domains at Week 4
Description: The DAS is a 4-point scale. The extent of functional impairment in 4 functional domains (dressing, hygiene, limb position and pain) was rated as follows: 0=no disability, 1=mild disability (noticeable but does not interfere significantly with normal activities), 2=moderate disability (normal activities require increased effort and/or assistance) and 3=severe disability (normal activities limited). The percentage of subjects with at least one grade reduction in DAS for each of the individual domains at Week 4 is reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Number; unit: percentage of subjects
Arm/Group | Total Dysport®
Number analyzed (Participants) | 254
percentage of subjects
  Hygiene - Cycle 1 | 40.9
  Hygiene - Cycle 2: number analyzed (Participants) | 229
  Hygiene - Cycle 2 | 45.4
  Hygiene - Cycle 3: number analyzed (Participants) | 175
  Hygiene - Cycle 3 | 44.6
  Hygiene - Cycle 4: number analyzed (Participants) | 81
  Hygiene - Cycle 4 | 46.9
  Dressing - Cycle 1 | 40.9
  Dressing - Cycle 2: number analyzed (Participants) | 229
  Dressing - Cycle 2 | 47.2
  Dressing - Cycle 3: number analyzed (Participants) | 175
  Dressing - Cycle 3 | 46.9
  Dressing - Cycle 4: number analyzed (Participants) | 81
  Dressing - Cycle 4 | 53.1
  Limb Position - Cycle 1 | 55.5
  Limb Position - Cycle 2: number analyzed (Participants) | 229
  Limb Position - Cycle 2 | 59.4
  Limb Position - Cycle 3: number analyzed (Participants) | 175
  Limb Position - Cycle 3 | 60.6
  Limb Position - Cycle 4: number analyzed (Participants) | 81
  Limb Position - Cycle 4 | 53.1
  Pain - Cycle 1 | 33.1
  Pain - Cycle 2: number analyzed (Participants) | 229
  Pain - Cycle 2 | 36.7
  Pain - Cycle 3: number analyzed (Participants) | 175
  Pain - Cycle 3 | 42.3
  Pain - Cycle 4: number analyzed (Participants) | 81
  Pain - Cycle 4 | 48.1

29. Secondary Outcome: Mean Change From Baseline to Week 4 for Angle of Arrest (XV1), Angle of Catch (XV3) and Angle of Spasticity (X) in Extrinsic Finger Flexors as PTMG
Description: The Tardieu Scale (TS) was used to measure spasticity in extrinsic finger flexors. The TS is administered by applying passive stretch to a muscle group at two velocities. Slow speed of muscle stretch measures the range of passive motion. During a slow stretching movement, the examiner determines the angle of movement arrest, either due to subject discomfort or a mechanical resistance. The same movement is repeated at high velocity (as fast as possible) to determine the angle of catch and release. The angle of movement arrest at slow velocity (XV1) and the angle of catch at fast speed (XV3) were recorded. The spasticity angle (X) was calculated as the difference between XV1 and XV3. Mean changes in Angles XV1, XV3 and X from baseline to Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Total Dysport®
Number analyzed (Participants) | 144
Degrees
  Angle of Spasticity (X) - Cycle 1 | -33.5 (54)
  Angle of Spasticity (X) - Cycle 2: number analyzed (Participants) | 133
  Angle of Spasticity (X) - Cycle 2 | -33.9 (55.9)
  Angle of Spasticity (X) - Cycle 3: number analyzed (Participants) | 98
  Angle of Spasticity (X) - Cycle 3 | -43.3 (57.8)
  Angle of Spasticity (X) - Cycle 4: number analyzed (Participants) | 56
  Angle of Spasticity (X) - Cycle 4 | -35.9 (48)
  Angle of Arrest (XV1) - Cycle 1 | 24.3 (36.1)
  Angle of Arrest (XV1) - Cycle 2: number analyzed (Participants) | 133
  Angle of Arrest (XV1) - Cycle 2 | 25.9 (36.5)
  Angle of Arrest (XV1) - Cycle 3: number analyzed (Participants) | 98
  Angle of Arrest (XV1) - Cycle 3 | 24.9 (38.7)
  Angle of Arrest (XV1) - Cycle 4: number analyzed (Participants) | 56
  Angle of Arrest (XV1) - Cycle 4 | 21.8 (39.6)
  Angle of Catch (XV3) - Cycle 1 | 57.8 (55.1)
  Angle of Catch (XV3) - Cycle 2: number analyzed (Participants) | 133
  Angle of Catch (XV3) - Cycle 2 | 59.8 (57.8)
  Angle of Catch (XV3) - Cycle 3: number analyzed (Participants) | 98
  Angle of Catch (XV3) - Cycle 3 | 68.2 (55.6)
  Angle of Catch (XV3) - Cycle 4: number analyzed (Participants) | 56
  Angle of Catch (XV3) - Cycle 4 | 57.7 (52.6)

30. Secondary Outcome: Mean Change From Baseline to Week 4 for Spasticity Grade (Y) in Extrinsic Finger Flexors as PTMG
Description: The TS was used to measure spasticity in extrinsic finger flexors. The TS is administered by applying passive stretch to a muscle group. The spasticity grade (Y) assesses quality of muscle reaction on a 5-point scale (measured at fast speed): 0 =No resistance throughout passive movement, 1=slight resistance throughout passive movement, 2=clear catch at precise angle, interrupting passive movement, followed by release, 3=fatigable clonus (less than 10 seconds when maintaining pressure) occurring at a precise angle, followed by release. 4=unfatigable clonus (more than 10 seconds when maintaining pressure) occurring at precise angle. Mean changes in spasticity grade (Y) from baseline to Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 144
units on a scale
  Cycle 1 | -0.6 (0.7)
  Cycle 2: number analyzed (Participants) | 133
  Cycle 2 | -0.6 (0.8)
  Cycle 3: number analyzed (Participants) | 98
  Cycle 3 | -0.6 (0.8)
  Cycle 4: number analyzed (Participants) | 56
  Cycle 4 | -0.5 (0.7)

31. Secondary Outcome: Mean Change From Baseline to Week 4 for Angle of Arrest (XV1), Angle of Catch (XV3) and Angle of Spasticity (X) in Elbow Flexors as PTMG
Description: The TS was used to measure spasticity in elbow flexors. The TS is administered by applying passive stretch to a muscle group at two velocities. Slow speed of muscle stretch measures the range of passive motion. During a slow stretching movement, the examiner determines the angle of movement arrest, either due to subject discomfort or a mechanical resistance. The same movement is repeated at high velocity (as fast as possible) to determine the angle of catch and release. The angle of movement arrest at slow velocity (XV1) and the angle of catch at fast speed (XV3) were recorded. The spasticity angle (X) was calculated as the difference between XV1 and XV3. Mean changes in Angles XV1, XV3 and X from baseline to Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Total Dysport®
Number analyzed (Participants) | 69
Degrees
  Angle of Spasticity (X) - Cycle 1 | -26.4 (24.9)
  Angle of Spasticity (X) -Cycle 2: number analyzed (Participants) | 59
  Angle of Spasticity (X) -Cycle 2 | -31 (27.7)
  Angle of Spasticity (X) -Cycle 3: number analyzed (Participants) | 42
  Angle of Spasticity (X) -Cycle 3 | -33.3 (26)
  Angle of Spasticity (X) -Cycle 4: number analyzed (Participants) | 14
  Angle of Spasticity (X) -Cycle 4 | -46.4 (17.3)
  Angle of Arrest (XV1) - Cycle 1 | -0.4 (14.9)
  Angle of Arrest (XV1) - Cycle 2: number analyzed (Participants) | 59
  Angle of Arrest (XV1) - Cycle 2 | 1.3 (13.3)
  Angle of arrest (XV1) - Cycle 3: number analyzed (Participants) | 42
  Angle of arrest (XV1) - Cycle 3 | 2.2 (10.6)
  Angle of Arrest (XV1) - Cycle 4: number analyzed (Participants) | 14
  Angle of Arrest (XV1) - Cycle 4 | -2.5 (9.4)
  Angle of Catch (XV3) - Cycle 1 | 26.0 (26.1)
  Angle of Catch (XV3) - Cycle 2: number analyzed (Participants) | 59
  Angle of Catch (XV3) - Cycle 2 | 32.3 (28.8)
  Angle of Catch (XV3) - Cycle 3: number analyzed (Participants) | 42
  Angle of Catch (XV3) - Cycle 3 | 35.5 (27.3)
  Angle of Catch (XV3) - Cycle 4: number analyzed (Participants) | 14
  Angle of Catch (XV3) - Cycle 4 | 43.9 (23.1)

32. Secondary Outcome: Mean Change From Baseline to Week 4 for Spasticity Grade (Y) in Elbow Flexors as PTMG
Description: The TS was used to measure spasticity in elbow flexors.The TS is administered by applying passive stretch to a muscle group. The spasticity grade (Y) assesses quality of muscle reaction on a 5-point scale (measured at fast speed): 0 =No resistance throughout passive movement, 1=slight resistance throughout passive movement, 2=clear catch at precise angle, interrupting passive movement, followed by release, 3=fatigable clonus (less than 10 seconds when maintaining pressure) occurring at a precise angle, followed by release. 4=unfatigable clonus (more than 10 seconds when maintaining pressure) occurring at precise angle. Mean changes in spasticity grade (Y) from baseline to Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 69
units on a scale
  Cycle 1 | -0.3 (0.5)
  Cycle 2: number analyzed (Participants) | 59
  Cycle 2 | -0.4 (0.7)
  Cycle 3: number analyzed (Participants) | 42
  Cycle 3 | -0.5 (0.7)
  Cycle 4: number analyzed (Participants) | 14
  Cycle 4 | -0.6 (0.5)

33. Secondary Outcome: Mean Change From Baseline to Week 4 for Angle of Arrest (XV1), Angle of Catch (XV3) and Angle of Spasticity (X) in Wrist Flexors as PTMG
Description: The TS was used to measure spasticity in wrist flexors. The TS is administered by applying passive stretch to a muscle group at two velocities. Slow speed of muscle stretch measures the range of passive motion. During a slow stretching movement, the examiner determines the angle of movement arrest, either due to subject discomfort or a mechanical resistance. The same movement is repeated at high velocity (as fast as possible) to determine the angle of catch and release. The angle of movement arrest at slow velocity (XV1) and the angle of catch at fast speed (XV3) were recorded. The spasticity angle (X) was calculated as the difference between XV1 and XV3. Mean changes in Angles XV1, XV3 and X from baseline to Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Total Dysport®
Number analyzed (Participants) | 39
Degrees
  Angle of Spasticity (X) - Cycle 1 | -23.3 (32.5)
  Angle of Spasticity (X) - Cycle 2: number analyzed (Participants) | 34
  Angle of Spasticity (X) - Cycle 2 | -28.8 (37.1)
  Angle of Spasticity (X) - Cycle 3: number analyzed (Participants) | 23
  Angle of Spasticity (X) - Cycle 3 | -21.7 (35.2)
  Angle of Spasticity (X) - Cycle 4: number analyzed (Participants) | 10
  Angle of Spasticity (X) - Cycle 4 | -13.5 (29.3)
  Angle of Arrest (XV1) - Cycle 1 | 12.6 (21.3)
  Angle of Arrest (XV1) - Cycle 2: number analyzed (Participants) | 34
  Angle of Arrest (XV1) - Cycle 2 | 16.4 (23.9)
  Angle of Arrest (XV1) - Cycle 3: number analyzed (Participants) | 23
  Angle of Arrest (XV1) - Cycle 3 | 18.6 (30.6)
  Angle of Arrest (XV1) - Cycle 4: number analyzed (Participants) | 10
  Angle of Arrest (XV1) - Cycle 4 | 19.0 (24.8)
  Angle of Catch (XV3) - Cycle 1 | 35.9 (35.0)
  Angle of Catch (XV3) - Cycle 2: number analyzed (Participants) | 34
  Angle of Catch (XV3) - Cycle 2 | 45.2 (37.7)
  Angle of Catch (XV3) - Cycle 3: number analyzed (Participants) | 23
  Angle of Catch (XV3) - Cycle 3 | 40.3 (33.3)
  Angle of Catch (XV3) - Cycle 4: number analyzed (Participants) | 10
  Angle of Catch (XV3) - Cycle 4 | 32.5 (28.1)

34. Secondary Outcome: Mean Change From Baseline to Week 4 for Spasticity Grade (Y) in Wrist Flexors as PTMG
Description: The TS was used to measure spasticity in wrist flexors. The TS is administered by applying passive stretch to a muscle group. The spasticity grade (Y) assesses quality of muscle reaction on a 5-point scale (measured at fast speed): 0 =No resistance throughout passive movement, 1=slight resistance throughout passive movement, 2=clear catch at precise angle, interrupting passive movement, followed by release, 3=fatigable clonus (less than 10 seconds when maintaining pressure) occurring at a precise angle, followed by release. 4=unfatigable clonus (more than 10 seconds when maintaining pressure) occurring at precise angle. Mean changes in spasticity grade (Y) from baseline to Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 39
units on a scale
  Cycle 1 | -0.7 (1.1)
  Cycle 2: number analyzed (Participants) | 34
  Cycle 2 | -0.9 (1.0)
  Cycle 3: number analyzed (Participants) | 23
  Cycle 3 | -0.6 (0.9)
  Cycle 4: number analyzed (Participants) | 10
  Cycle 4 | -0.3 (0.7)

35. Secondary Outcome: Mean Change From Baseline to Week 4 for Angle of Arrest (XV1), Angle of Catch (XV3) and Angle of Spasticity (X) in Shoulder Extensors
Description: The TS was used to measure spasticity in shoulder extensors. The TS is administered by applying passive stretch to a muscle group at two velocities. Slow speed of muscle stretch measures the range of passive motion. During a slow stretching movement, the examiner determines the angle of movement arrest, either due to subject discomfort or a mechanical resistance. The same movement is repeated at high velocity (as fast as possible) to determine the angle of catch and release. The angle of movement arrest at slow velocity (XV1) and the angle of catch at fast speed (XV3) were recorded. The spasticity angle (X) was calculated as the difference between XV1 and XV3. Mean changes in Angles XV1, XV3 and X from baseline to Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Total Dysport®
Number analyzed (Participants) | 67
Degrees
  Angle of Spasticity (X) - Cycle 1: number analyzed (Participants) | 35
  Angle of Spasticity (X) - Cycle 1 | -13.3 (24.6)
  Angle of Spasticity (X) - Cycle 2 | -10.8 (30.1)
  Angle of Spasticity (X) - Cycle 3: number analyzed (Participants) | 55
  Angle of Spasticity (X) - Cycle 3 | -6.4 (23.5)
  Angle of Spasticity (X) - Cycle 4: number analyzed (Participants) | 32
  Angle of Spasticity (X) - Cycle 4 | -7.2 (27.4)
  Angle of Arrest (XV1) - Cycle 1: number analyzed (Participants) | 35
  Angle of Arrest (XV1) - Cycle 1 | 7.2 (16.0)
  Angle of Arrest (XV1) - Cycle 2 | 6.4 (23.0)
  Angle of Arrest (XV1) - Cycle 3: number analyzed (Participants) | 55
  Angle of Arrest (XV1) - Cycle 3 | 10.7 (23.8)
  Angle of Arrest (XV1) - Cycle 4: number analyzed (Participants) | 32
  Angle of Arrest (XV1) - Cycle 4 | 10.8 (26.1)
  Angle of Catch (XV3) - Cycle 1: number analyzed (Participants) | 35
  Angle of Catch (XV3) - Cycle 1 | 20.5 (22.7)
  Angle of Catch (XV3) - Cycle 2 | 17.2 (26.9)
  Angle of Catch (XV3) - Cycle 3: number analyzed (Participants) | 55
  Angle of Catch (XV3) - Cycle 3 | 17.1 (24.5)
  Angle of Catch (XV3) - Cycle 4: number analyzed (Participants) | 32
  Angle of Catch (XV3) - Cycle 4 | 18.0 (19.6)

36. Secondary Outcome: Mean Change From Baseline to Week 4 for Spasticity Grade (Y) in Shoulder Extensors
Description: The TS was used to measure spasticity in shoulder extensors. The TS is administered by applying passive stretch to a muscle group. The spasticity grade (Y) assesses quality of muscle reaction on a 5-point scale (measured at fast speed): 0 =No resistance throughout passive movement, 1=slight resistance throughout passive movement, 2=clear catch at precise angle, interrupting passive movement, followed by release, 3=fatigable clonus (less than 10 seconds when maintaining pressure) occurring at a precise angle, followed by release. 4=unfatigable clonus (more than 10 seconds when maintaining pressure) occurring at precise angle. Mean changes in spasticity grade (Y) from baseline to Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 67
units on a scale
  Cycle 1: number analyzed (Participants) | 35
  Cycle 1 | -0.1 (0.4)
  Cycle 2 | -0.1 (0.6)
  Cycle 3: number analyzed (Participants) | 55
  Cycle 3 | -0.2 (0.7)
  Cycle 4: number analyzed (Participants) | 32
  Cycle 4 | -0.2 (0.5)

37. Secondary Outcome: Mean Change From Baseline in Active Range of Motion (AROM) at Week 4 in the 3 Possible PTMGs
Description: The AROM was assessed by the range of extension achieved by the subject moving each joint in the PTMGs (extrinsic finger flexors, elbow flexors and wrist flexors) without assistance. A goniometer was used for measurements in the elbow and wrist flexors but not for measurements in the extrinsic finger flexors. Mean changes in AROM in the 3 possible PTMGs from baseline to Week 4 are reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 144
units on a scale
  Extrinsic Finger Flexors: Cycle 1 | 31.3 (40.9)
  Extrinsic Finger Flexors: Cycle 2: number analyzed (Participants) | 133
  Extrinsic Finger Flexors: Cycle 2 | 34.4 (45)
  Extrinsic Finger Flexors: Cycle 3: number analyzed (Participants) | 98
  Extrinsic Finger Flexors: Cycle 3 | 33.5 (47.1)
  Extrinsic Finger Flexors: Cycle 4: number analyzed (Participants) | 56
  Extrinsic Finger Flexors: Cycle 4 | 38 (53.4)
  Elbow Flexors: Cycle 1: number analyzed (Participants) | 69
  Elbow Flexors: Cycle 1 | 10.7 (25.5)
  Elbow Flexors: Cycle 2: number analyzed (Participants) | 59
  Elbow Flexors: Cycle 2 | 17.6 (23.3)
  Elbow Flexors: Cycle 3: number analyzed (Participants) | 42
  Elbow Flexors: Cycle 3 | 14.5 (24.1)
  Elbow Flexors: Cycle 4: number analyzed (Participants) | 14
  Elbow Flexors: Cycle 4 | 13.6 (20.6)
  Wrist Flexors: Cycle 1: number analyzed (Participants) | 39
  Wrist Flexors: Cycle 1 | 17.3 (28.6)
  Wrist Flexors: Cycle 2: number analyzed (Participants) | 34
  Wrist Flexors: Cycle 2 | 23 (32.7)
  Wrist Flexors: Cycle 3: number analyzed (Participants) | 23
  Wrist Flexors: Cycle 3 | 22 (30.9)
  Wrist Flexors: Cycle 4: number analyzed (Participants) | 10
  Wrist Flexors: Cycle 4 | 3 (25.1)

38. Secondary Outcome: Mean Change From Baseline at Week 4 in Ease of Applying a Splint
Description: The ease of applying a splint was evaluated on a 6-point scale (0= no splint needed, -1= splint needed and applied with no difficulty, -2= splint needed and applied with mild difficulty, -3= splint needed and applied with moderate difficulty, -4= splint needed and applied with severe difficulty, -5= splint needed,but unable to apply). Mean change in ease of applying a splint from baseline to Week 4 was reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 218
units on a scale
  Cycle 1 | -0.4 (1.1)
  Cycle 2: number analyzed (Participants) | 196
  Cycle 2 | -0.4 (1.3)
  Cycle 3: number analyzed (Participants) | 137
  Cycle 3 | -0.4 (1.4)
  Cycle 4: number analyzed (Participants) | 56
  Cycle 4 | -0.4 (1)

39. Secondary Outcome: Mean Change From Baseline in Modified Frenchay Scale (MFS) at Week 4
Description: The MFS was used to measure upper limb active function. Each subject was video taped while performing specific tasks. The videos were sent to a central provider and were read and scored by two independent readers blinded to the timing of the video and to treatment. These central assessments were used for the analysis of efficacy endpoints. The MFS consists of 10 tasks asking the subject to reach, grasp, carry and release different objects of different sizes which subjects are likely to use in their daily life. Each of these tasks was rated on a 10 point scale ranging from no movement to normal movement; for each task, the score 5 is used to rate a task barely accomplished. Mean change in MFS from baseline to Week 4 was reported.
Time Frame: At Week 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 219
units on a scale
  Cycle 1 | 0.4 (0.77)
  Cycle 2: number analyzed (Participants) | 190
  Cycle 2 | 0.51 (0.8)
  Cycle 3: number analyzed (Participants) | 138
  Cycle 3 | 0.44 (0.82)
  Cycle 4: number analyzed (Participants) | 56
  Cycle 4 | 0.4 (0.75)

40. Secondary Outcome: Mean Change From Baseline in Short Form (36) Health Survey (SF-36) Quality of Life (QoL) at End of Study/Early Withdrawal Visit
Description: Subjects were asked to complete the SF-36 questionnaires prior to the study treatment at baseline and at the end of study/early withdrawal visit. The SF-36 is a generic non-preference based health status measure. This instrument assessed subject health across 8 variable dimensions, which are specific health domains such as physical functioning, social functioning and vitality. Each variable item score is coded and turned into a 0-100 scale where 0 indicates the worst and 100 indicates the best possible health state for both the Physical Component Summary (PCS) and Mental Component Summary (MCS) of the questionnaire. Baseline results and the change from baseline to end of study/early withdrawal for the PCS and MCS are reported.
Time Frame: Up to Week 52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 244
units on a scale
  PCS Baseline | 37.49 (8.94)
  PCS Change: number analyzed (Participants) | 229
  PCS Change | 1.07 (6.76)
  MCS Baseline | 46.88 (13.09)
  MCS Change: number analyzed (Participants) | 229
  MCS Change | 0.96 (11.11)

41. Secondary Outcome: Mean Change From Baseline in European 5 Dimensions, 5 Level (EQ-5D-5L) QoL at End of Study/Early Withdrawal Visit
Description: Subjects were asked to complete the EQ-5D-5L QoL questionnaires prior to the study treatment at baseline and at the end of study/early withdrawal visit. The EQ-5D-5L index is a generic preference based measure of health related QoL producing utility scores that represent subject preferences for particular health states. This instrument rated subject health state looking at 5 specific dimensions such as mobility, self-care, usual activity, pain/discomfort and anxiety/depression and scored their general health state. Each dimension has 5 levels of severity (no problems, slight problems,moderate problems, severe problems and extreme problems). In addition, a visual analogue scale (VAS) ranging from 0 to 100 was also included for the patients to summarize their overall health status, where 0 is the worst and 100 the best possible health state. The mean values for each dimension and the VAS scores at baseline and at the end of-study /early withdrawal are reported.
Time Frame: Up to Week 52
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 249
units on a scale
  Anxiety/Depression Baseline | 1.9 (0.9)
  Anxiety/Depression Change: number analyzed (Participants) | 231
  Anxiety/Depression Change | -0.1 (0.9)
  Mobility Baseline | 2.8 (0.9)
  Mobility Change: number analyzed (Participants) | 231
  Mobility Change | 0 (0.8)
  Pain/Discomfort Baseline | 2.1 (1)
  Pain/Discomfort Change: number analyzed (Participants) | 231
  Pain/Discomfort Change | -0.2 (0.9)
  Self-Care Baseline | 2.4 (1)
  Self-Care Change: number analyzed (Participants) | 231
  Self-Care Change | 0 (0.8)
  Usual Activities Baseline | 2.8 (1)
  Usual Activities Change: number analyzed (Participants) | 231
  Usual Activities Change | -0.2 (1)
  VAS Baseline | 63.6 (19.7)
  VAS Change: number analyzed (Participants) | 231
  VAS Change | 2.8 (19)

ADVERSE EVENTS:
Time Frame: Up to Week 52
Description: An AE was reported as emergent if it arose (i.e. started or worsened in severity) in the treatment phase after the subject received study medication.
Arm/Group | Total Dysport®
Serious Adverse Events (participants affected / at risk) | 21/254
Other Adverse Events (participants affected / at risk) | 142/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Dysport® (N=254)
Haematoma (Vascular disorders) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Death
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Device malfunction (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Affect lability (Psychiatric disorders) | 1 (1)
Affective disorder (Psychiatric disorders) | 1 (1)
Mania (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) — Death
Myocardial infarction (Cardiac disorders) | 1 (1) — Death
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (2)
Brain injury (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Dysport® (N=254)
Hypertension (Vascular disorders) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 20 (25)
Hand fracture (Injury, poisoning and procedural complications) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 4 (4)
Humerus fracture (Injury, poisoning and procedural complications) | 3 (3)
Alanine aminotransferase increased (Investigations) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Seasonal allergy (Immune system disorders) | 3 (3)
Headache (Nervous system disorders) | 6 (6)
Epilepsy (Nervous system disorders) | 3 (6)
Paraesthesia (Nervous system disorders) | 3 (3)
Asthenia (General disorders) | 5 (5)
Fatigue (General disorders) | 7 (8)
Pyrexia (General disorders) | 3 (5)
Peripheral swelling (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 4 (4)
Injection site bruising (General disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 5 (5)
Depression (Psychiatric disorders) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (18)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 13 (14)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bronchitis (Infections and infestations) | 5 (5)
Nasopharyngitis (Infections and infestations) | 6 (7)
Urinary tract infection (Infections and infestations) | 6 (10)
Influenza (Infections and infestations) | 4 (4)
Sinusitis (Infections and infestations) | 4 (4)
Cystitis (Infections and infestations) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 3 (3)
Herpes zoster (Infections and infestations) | 3 (3)
Upper respiratory tract (Infections and infestations) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No